CLINICAL TRIAL: NCT05300815
Title: Identifying Which Adverse Events Associated With Dry Needling Should be Included For Informed Consent: A Modified e-Delphi Study
Status: Completed | Type: Observational
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Edmund Ickert, Primary Investigator, Youngstown State University
Other Study IDs: 2022-117
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Dry Needling
Keywords: informed consent; adverse event; delphi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dry Needling Experts: Experts will be defined as adult individuals with a high level of knowledge within the area of patient safety and adverse events related to dry needling which will be confirmed using the following eligibility criteria:
  (1) Must have >= 5 years of clinical practice performing dry needling and at least ONE of the following secondary criteria:
  1. Certification in Dry Needling
  2. Completion of a manual therapy fellowship that included dry needling training
  3. >= 1 total scholarly product (poster presentation, author of a peer-reviewed publication) involving the use of dry needling
  Eligible participants will be identified through existing professional networks and social media/internet-based searching. They will be recruited worldwide and be aged 18 or above, able to read and write in English, and willing to provide signed informed consent.
  Interventions: Other: Delphi Questionaire

INTERVENTIONS:
Other: Delphi Questionaire — This study involves the use of questionnaires across 3 rounds as follows:
  The objectives of round 1 are to collect participant demographic information and generate a list of adverse events. Round 1 will be open for 3 weeks with email reminders being provided at weeks 1 and 2.
  The objectives of round 2 will be to share a list of adverse events generated from round 1 (with the addition of adverse events identified in literature if not generated in round 1) and allow participants to rate from 1-4 how important each item is for inclusion on informed consent. As per round 1, the round 2 questionnaire will remain active for 3 weeks with email reminders sent at weeks 1 and 2.
  The objective of round 3 is to further gain consensus on adverse events from the results of round 2 where agreement was not reached. Round 3 remains active for 3 weeks with email reminders sent at weeks 1 and 2.

SUMMARY:
Dry Needling is an intervention that continues to gain widespread interest as a treatment adjunct for various pathological conditions. With the increased use of dry needling in the clinic, there comes a need for additional research to investigate the adverse events associated with the use of dry needling. Informed Consent is a process that is legally required in many states prior to the performance of a treatment intervention like dry needling. It is important therefore to identify which of these adverse events should be included in an informed consent process.

DETAILED DESCRIPTION:
Over the past 10 years, there have been a great deal of studies that examined the application of DN to varying pathological conditions. Some of the more recent studies involving the application of DN for various conditions include: temporomandibular joint dysfunction (TMD), post-stroke, plantar heel pain or plantar fasciitis, osteoarthritis, headache, fibromyalgia, neck and shoulder pain, lateral epicondylagia, back pain, and hallux valgus. In addition to studies that applied DN to specific pathological conditions, the effects of DN have also been studied. DN has been shown to: improve spasticity and range of motion (ROM), improve flexibility of muscles, myofascial trigger point pain, scar tissue, and neuromuscular control.

As DN interest continues to expand and studies continue to show the feasibility of applying DN to a wider range of pathological conditions, there is a need to understand the risks related to the use of DN. Understanding the risks associated with DN will allow for improvements in clinical decision making regarding whether DN is an appropriate choice for the patient. Informed Consent (IC) is a means of respecting the autonomous preferences of persons seeking health care or participation in research. One of the important elements of IC is the need to be explicit and descriptive about the risks of treatment which include: the nature of the risk, the probability the risk will occur, the severity of the risk, and the proximity of the risk. These are important elements that would allow the patient to be able to consider the risks to benefit ratio of a given intervention and will lead to making a better informed decision regarding their own care. Without the risks being properly identified for the intervention, the IC process could not be adhered to and the patient would not be able to make a well-informed decision regarding their own care.

There have been no studies that have described how the risks associated with DN should be incorporated during the IC process to drive patient-centered care and autonomy in decision making. The purpose of this study will be to utilize a Modified Delphi framework to identify expert consensus on which risks should be included in the IC process.

ELIGIBILITY:
Inclusion Criteria:

Physical Therapists who:

Have >= 7 years of clinical practice performing dry needling and at least ONE of the following secondary criteria:

1. Certification in Dry Needling
2. Completion of a manual therapy fellowship that included dry needling training
3. >= 1 total scholarly product (poster presentation, author of a peer-reviewed publication)

Exclusion Criteria:

* Not a Physical Therapist
* Has less than 7 years experience in dry needling
* Does not meet the secondary criteria established in the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical Therapists who have >= 7 years of experience performing dry needling and at least ONE of the following secondary criteria:
  1. Certification in Dry Needling
  2. Completion of a manual therapy fellowship that included dry needling training
  3. >= 1 total scholarly product (poster presentation, author of a peer-reviewed publication)
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | Baseline
  Contains questions about the characteristics of the participants
Round 1 Questionnaire | Baseline to 3 weeks
  Participants list known adverse events associated with dry needling
Round 2 Questionnaire | 3 weeks to 6 weeks
  Participants identify which adverse events they agree should be included during informed consent.
Round 3 Questionnaire | 6 weeks to 9 weeks
  Participants will see the results from round 2 and further identify which adverse events should be included for informed consent.

CONTACTS AND LOCATIONS:
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funabashi M, Pohlman KA, Gorrell LM, Salsbury SA, Bergna A, Heneghan NR. Expert consensus on a standardised definition and severity classification for adverse events associated with spinal and peripheral joint manipulation and mobilisation: protocol for an international e-Delphi study. BMJ Open. 2021 Nov 11;11(11):e050219. doi: 10.1136/bmjopen-2021-050219. PMID 34764170